CLINICAL TRIAL: NCT03620682
Title: Using Smartphone Technology to Provide Mental Health Interventions for Homeless Youth
Brief Title: Homeless Youth Study - Stepping Stone Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Alyson Zalta, Assistant Professor, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14112402
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile mental health intervention (Experimental): Participants will receive emotional support and problem-solving / stress-management skills via over-the-phone coaching sessions and mobile applications.
  Interventions: Behavioral: Coaching sessions; Behavioral: Mobile applications

INTERVENTIONS:
Behavioral: Coaching sessions — Participants receive three 30-minute phone sessions with a doctorate-level therapist over the course of one month. These sessions are skills-based and focus on improving participants' problem solving through cognitive-behavioral techniques. Participants are allowed to text the therapist between sessions for information and support.
Behavioral: Mobile applications — Participants will have access to 3 mobile apps for the duration of the study, and after it ends. One app will push participants a daily, self-reflective survey to complete, and a daily motivational or instructional tip to rate. Other apps will provide education and exercises on various aspects of mental health and wellness, such as sleep and relaxation.

SUMMARY:
Homelessness is associated with a multitude of negative consequences including an increased risk for mental health problems. Once homeless, these individuals face significant barriers to mental health care and are therefore less likely to receive the treatment they need. Mobile technology may offer a novel platform for increasing access to mental health care in this population. Thus, the primary goals of this pilot study are to (1) establish the feasibility and acceptability of delivering a brief cognitive-behavioral intervention to homeless youth via smartphone technology, (2) examine the extent to which brief cognitive-behavioral interventions delivered via mobile technology improve mental health and trauma-related psychological symptoms in homeless youth, and (3) establish smartphone usage patterns among homeless youth to inform future interventions.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Homeless as defined by lacking "a fixed, regular, and adequate nighttime residence," (Department of Education) including youth who temporarily share the housing of others due to financial hardship
* Currently sleeping in a Chicago-based shelter (at least 50% of nights in the past week)
* Willingness and ability to comply with requirements of the study protocol

Exclusion Criteria:

* Involvement in risky behaviors that could interfere with the ability to fully engage in the study, as determined by the Principal Investigator
* Current involvement in legal proceedings
* Mental retardation or significant cognitive impairment
* Significant suicidal ideation indicated by a BDI-II item 9 score ≥ 2 or enacted suicidal behaviors within 6 months prior to eligibility
* Any concurrent psychotherapy of any duration
* Inability to understand study procedures and participate in the informed consent process

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | Baseline (week 0) to Endpoint (week 4)
  Adherence will be assessed based on number of coaching sessions attended over the course of the 1 month treatment period (range of 0 to 3).
Treatment satisfaction | Treatment endpoint (week 4)
  Participants will be asked to report the extent to which they were satisfied with the study, the extent to which they thought the study was helpful, and whether they would recommend the study to someone else. These responses are recorded on 5-point likert type scales with higher ratings indicating higher satisfaction.

SECONDARY OUTCOMES:
Depression symptoms | Baseline (week 0) to Endpoint (week 4)
  Depression symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The range is from 0-27. Higher values represent worse depression symptoms.
Posttraumatic Stress Disorder symptoms | Baseline (week 0) to Endpoint (week 4)
  PTSD symptoms will be assessed using the PTSD Checklist for DSM-5 (PCL-5). The range is from 0-80. Higher values represent worse PTSD symptoms.
Emotion Regulation | Baseline (week 0) to Endpoint (week 4)
  Ability to regulate emotion will be assessed using the Difficulties in Emotion Regulation Scale (DERS). Range is from 36 to 180. Higher scores suggest greater problems with emotion regulation.
Anxiety symptoms | Baseline (week 0) to Endpoint (week 4)
  Current symptoms of anxiety will be assessed using the State Anxiety scale of the State Trait Anxiety Inventory. Scores range from 20 to 80. Higher scores indicate greater anxiety.
Risky sexual behavior and substance use | Baseline (week 0) to Endpoint (week 4)
  Risky sexual behaviors and substance use will be assessed using the Centers for Disease Control and Prevention's Youth Risk Behavior Survey (2011).
Acceptability of treatment components | Endpoint (week 4)
  At the end of the treatment period, participants will rate the extent to which they liked each of the different treatment components (coaching sessions, text messages, apps, tips). Participants will also be asked to report the extent to which they used the skills that they learned in the coaching sessions.

OTHER OUTCOMES:
Acceptability of mental health treatment | Baseline (week 0) to Endpoint (week 4)
  Attitudes toward the mental health system will be assessed using an author-developed measure.
Positive and negative affect | Baseline (week 0) to Endpoint (week 4)
  Current positive and negative emotions will be assessed using the Positive and Negative Affect Schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson K Zalta, PhD, Principal Investigator — Rush University Medical Center

REFERENCES:
- [Derived] Schueller SM, Glover AC, Rufa AK, Dowdle CL, Gross GD, Karnik NS, Zalta AK. A Mobile Phone-Based Intervention to Improve Mental Health Among Homeless Young Adults: Pilot Feasibility Trial. JMIR Mhealth Uhealth. 2019 Jul 2;7(7):e12347. doi: 10.2196/12347. PMID 31267980

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT03620682/Prot_SAP_000.pdf